CLINICAL TRIAL: NCT03741283
Title: Optimisation of Nutrition and Medication for Acutely Admitted Older Medical Patients
Acronym: OptiNAM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Clinical Research Centre (Unknown); Region Hovedstadens Apotek (Other Government); Udviklings- og forskningspuljen, Danske Regioner og Sundhedskartellet (Unknown); Region Capital Denmark (Other); Regionernes Lægemiddelorganisation (Unknown)
Responsible Party: Principal Investigator, Ove Andersen, Head of Clinical Research Centre, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OptiNAM; VD-2018-390 -"optiNAM" (Other: Danish Data Protection Agency)
Record Dates: First submitted 2018-11-05; First posted 2018-11-14 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Aging; Malnutrition; Drug Prescribing
Keywords: Medicines optimisation; Multimodal interventions; Inflammation; Emergency Service, Hospital; Pharmacogenetics; Renal function; Food intake; Quality of life; Polypharmacy
MeSH Terms: conditions — Malnutrition; Inflammation; Emergencies | interventions — Dosage Forms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Optimisation of nutrition and medication (Experimental): N=approx.
  65 acutely admitted older medical patients with undernutrition or risk of undernutrition, and 35 without undernutrition or risk of undernutrition.
  Interventions: Other: Optimisation of nutrition and medication
- Standard care (No Intervention): N= approx. 65 acutely admitted older medical patients with undernutrition or risk of undernutrition, and 35 without undernutrition or risk of undernutrition.

INTERVENTIONS:
Other: Optimisation of nutrition and medication — 1. Inter-professional optimisation of medication prescribing:
     Study participants in the intervention group receives optimisation of medication prescribing at admission day (baseline) regardless of nutritional state. The intervention is performed in cooperation between a clinical pharmacist and a medical physician.
  2. Nutritional intervention:
  If positive screening for malnutrition or risk of malnutrition a dietetic intervention is initiated and if positive screening below interventions are initiated:
  * Dysphagia: occupational therapy intervention.
  * Oral cavity problems: odontological intervention.
  * Depression: geriatric intervention.
  * Low ADL: occupational therapy intervention and if positive screening for poor muscle strength: physiotherapeutic intervention.
  Arms: Optimisation of nutrition and medication

SUMMARY:
Malnutrition and inappropriate medication prescribing are highly prevalent among acutely admitted older medical patients leading to re-admissions, frailty, poor physical, performance compromised quality of life and mortality. Thus, the aim of this study is to optimise the nutrition and medication in older medical patients admitted to an acute care department at admission and up to 16 weeks after discharge. Participants in the intervention group receives a medication review and participants with malnutrition or risk of malnutrition additionally receive a transitional multimodal intervention. The control group receives standard care.

DETAILED DESCRIPTION:
The OptiNAM study is designed as a single-blinded randomised controlled trial starting upon admission and continues till 16 weeks after discharge. The trial has five sub-studies with three independent primary endpoints, all with individual sample size calculations.

The study consists of an intervention group and a control group. The control group receives standard care.

Patients that meet all inclusion criteria and none of the exclusion criteria are invited to participate. After signing a written informed consent, the participants are block randomised to either the intervention or control group.

The intervention group receives a personalised rehabilitation program, which is described below. Outcome measures are performed at baseline, week 8 and week 16 after after discharge, cf. section regarding outcome measures.

Sub study 1, Malnutrition:

As malnutrition among older patients has multifactorial etiology sub-study 1 investigates the effects of a multimodal transitional intervention on quality of life in acutely admitted older patients with malnutrition or risk of malnutrition (according to the Mini Nutritional Assessment - Short Form) from baseline (admission day) and 16 weeks after discharge compared to standard care. The intervention includes a medication review (cf. sub-study 2), a dietetic intervention and if clinical relevant physiotherapeutic-, occupational-, geriatric- and/or odontological intervention. It is secondary hypothesised that a multimodal intervention compared to standard care may improve the quality of life, nutritional status, energy- and protein intake, symptoms which compromise nutritional intake, physical performance, cognitive function, frailty, re-admissions, inflammation and biomarkers. A cost-benefit analysis will be conducted.

Dietetic intervention: The study subjects receives a personal diet plan during admission. The diet plan is reviewed at discharge by a dietician. To ensure optimal energy- and protein intake after discharge, a community-based dietician visit the participants for one hour in week 1, 2, 4 and 8.

Physiotherapeutic intervention: Participants with low ability to perform groceries shopping, cooking and/or eating are offered a community-based strength, balance and endurance training after discharge if they also have low muscle strength in the lower extremities. The training sessions are based on algorithms, have a duration of one hour, and are offered twice a week for 16 weeks after discharge.

Occupational intervention, Dysphagia: If relevant (EAT-10 score >=3), a hospital-based occupational therapist review and treat the dysphagia based on the Facial Oral Tract Therapy (FOTT) principle during admission. During the first week after discharge a community-based occupational therapist continues with the treatment. A maximum of two weekly visits of one hour throughout the interventions period is offered.

Occupational Intervention, low Ability to perform Activities of Daily Living (ADL): If the participant has low ability to perform grocery shopping, cooking and eating (evaluated by Functional Recovery Score <=2) then a community-based occupational therapist visit the participant during the first two weeks after discharge to evaluate the quality of activities of daily living. If relevant, and if there is a rehabilitation potential, seven visits of one hour is offered during the 16 weeks after discharge.

Geriatric intervention: If relevant (a Mini Geriatric Depression Score >=2), a geriatric physician conducts a clinical assessment of depression during admission and initiate treatment if necessary.

Odontological intervention: If relevant (participant reported pain in mouth, difficulties chewing or xerostomia), a dentist evaluate the dental status and oral health during admission, and if necessary encourage the participant to consult a dentist after discharge. If a participant shows insufficient oral hygiene a dental hygienist visits the participant after discharge twice during after discharge.

Sub-study 2, Medication optimisation:

Medication prescription for older patients is challenging and may be attributed to marked inter-individual variations in general health, comorbidities, organ function, pharmacokinetic and pharmacodynamic properties, biological age and physical performance. Thus, the "one size fits all" approach is probably inappropriate in older patients. The aim of sub-study 2 is to investigate the investigate the effect of an inter-professional conducted medication review during admission in an acute care department regardless of the nutritional status in the study participant, thus all subjects in the intervention group receive a medication review. It is hypothesized that inter-professional conducted medication reviews reduce the Medication Appropriateness Index score (MAI score) in the intervention group eight weeks after discharge compared to the control group. It is secondary hypothesized that inter-professional conducted medication reviews improve: lack of medication prescribing for a condition/disease, inappropriate polypharmacy and suboptimal medication prescribing of high risk medications.

Sub-study 3, Accuracy of renal function estimates and the consequence for prescribing recommendations guidelines:

Accuracy in renal function estimates is essential for optimization of medication prescribing since 40 % of all medication or their active metabolites is renally excreted. Lack of medication prescribing and dose adjustment according to the renal function is common in older patients with renal impairment and can result in overdosing, adverse drug reactions, hospital admissions, reduced quality of life and mortality. The gold standard for measuring glomerular filtration rate (GFR) is an exogenous filtration marker. However, this method is costly, time consuming and thus impractical in a clinical setting. Therefore, GFR is often estimated on serum concentrations of an endogen biomarker. Sub-study 3 aim to investigate which biomarker(s) and equation most accurately estimate the GFR in older medical patients who have been acutely admitted.

Sub-study 4, Pharmacogenetic test on cytochrome 450 variations and its potential for optimization of medication prescribing:

Cytochrome 450 enzymes are responsible for metabolism of up to 80% of all medications. The enzyme complex is mainly found in liver but are also present in intestinal mucosa, skin, lungs, brain and kidneys. There are major genetic inter-individual differences in the activity of the CYP 450 complex, resulting in lack of therapeutic effects, lack of effect or adverse drug reactions. Insight into these genetic inter-individual differences via pharmacogenetic tests possess a potential in optimization of medication prescribing with regard to therapeutic effects, compliance and risk of side effects. Thus, sub-study 4 wish to descriptively investigate the potential of pharmacogenetic test on cytochrome 450 variations.

Sub-study 5, Assessment of Frailty:

Frailty is a common clinical syndrome in older adults and defined as state of increased vulnerability resulting from decline in reserve capacity and function across multiple physiologic systems. Frailty affects the person's ability to cope with everyday life and leads to high risk for falls, disability, hospitalization and mortality. The frailty assessment is based on two different frailty scoring systems, Frieds "Frailty Phenotype" and Morley's "Frail Scale", examined at admission and 8 and 16 weeks after discharge. The purpose of the assessment is to evaluate which frailty measure is the best applicable in describing the patients and changes in their functional level. As there is no gold standard we use FI-Outref as an independent measure of frailty. FI-OutRef is a Frailty Index, based on standard admission laboratory test results Outside of the Reference interval.

ELIGIBILITY:
Inclusion Criteria:

* ≥65 years
* Acutely admitted medical patients
* Understand and speak Danish
* Caucasian
* Resident in Municipality: Brøndby, Hvidovre or Copenhagen

Exclusion Criteria:

* Unable to cooperate cognitively
* Terminal/suicidal patients
* Patients in isolation

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 193 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2022-07-15 (Estimated); Study Completion 2022-07-15 (Estimated)

PRIMARY OUTCOMES:
Changes in quality of life score EuroQol- 5 Dimensions- 5 Levels (sub-study 1) | Baseline (admission day), week 8 and week 16.
  Patient administered quality of life scoring system with focus on mobility, daily activities, pain and discomfort and depression.
Changes in Medication Appropriateness Index-score" (sub-study 2) | Baseline (admission day), week 8 and week 16.
  Medical physician, geriatric or senior pharmacist perform the MAI-scoring to evaluate the appropriateness of the medication prescribing.
Accuracy of renal function estimates (sub-study 3) - cystatin C | Baseline (admission day) or no later than 14 days after admission
  Differences between GFR measured by a renally excreted radioactive labeled isotope (chromium 51-Cr-EDTA or 99mTc diethylenetriaminepentaacetic acid) and estimated GFR based on Creatinine and Cystatin C or a combination of the biomarkers.

SECONDARY OUTCOMES:
Walking speed to evaluate the development in physical performance | Baseline (admission day), week 8 and week 16.
  4-Meter Walk Test
Functional measurement to evaluate the development in physical performance | Baseline (admission day), week 8 and week 16.
  30-second chair stand test
Functional measurement to evaluate the development in physical performance | Baseline (admission day), week 8 and week 16.
  handgrip strength test
Functional measurement to evaluate the development in physical performance | Baseline (admission day), week 8 and week 16.
  The de morton mobility index
Measure of physically active time and number of steps taken | Week 1, week 8 and week 16 after discharge
  Assessed by applying an activPAL chip to the thigh for one week
Frailty assessment | Baseline (admission day), week 8 and week 16.
  Fried frailty phenotype
Frailty assessment | Baseline (admission day), week 8 and week 16.
  Morleys frail questionnaire
Anthropometric measurement to monitor changes in bodyweight | Baseline (admission day), week 8 and week 16.
  Bodyweight
Cognitive test aiming to evaluate cognitive function | Baseline (admission day), week 8 and week 16
  Orientation Memory Concentration test
Patient records | Baseline (admission day), week 8 and week 16.
  Contacts related to the health care system, medication lists, use of municipal services
Standard admission blood work | Baseline (admission day), week 8 and week 16.
  ALAT, albumin, alkaline phosphatase, bilirubin, CO2, CRP, haemoglobin, INR, K+, blood urea nitrogen, coagulation factors, leucocytes, neutrophils, MCH, MCV, Na+, thrombocytes, lactate-dehydrogenases, NGAL, β-trace protein and β-trace microglobulins.
Quality of life score, WHO-5 | Baseline (admission day), week 8 and week 16
  Patient administered quality of life scoring system with focus on general well-being on a scale from 0-100.
Cognitive performance | Week 8 and week 16
  Mini mental state examination
Cognitive performance | Week 8 and week 16
  Hopkins verbal learning test
Cognitive performance | Week 8 and week 16
  Trail making test
Cognitive performance | Week 8 and week 16
  Digit Symbol Substitution test
Assessment of dietary intake after admission | Week 8 and week 16
  24 hours dietary recall
Evaluation of medication under-prescribing | Baseline (admission day), week 8 and week 16
  Assessment of underutilization Index (AOU)
Inflammatory marker to evaluate the inflammatory state | Baseline (admission day), week 8 and week 16.
  SuPAR
Polypharmacy | Baseline (admission day), week 8 and week 16.
  The number of patients in polypharmacy
Potentially inappropriate medication to elderly | Baseline (admission day), week 8 and week 16.
  The number of potentially inappropriate medication prescriptions
Acceptance of suggested changes in medications | Baseline (admission day), week 8 and week 16.
  Frequency of physicians' acceptance of suggested changes in medications
Accuracy of renal function estimates - all biomarkers | Baseline (admission day) or no later than 14 days after admission.
  Differences between GFR measured by a renally excreted radioactive labeled isotope (chromium 51-Cr-EDTA or 99mTc diethylenetriaminepentaacetic acid) and estimated GFR based on Creatinine, Cystatin C, Beta-trace protein, Beta-2 microglobulin or a combination of the biomarkers.
Dosing discrepancies of renal risk medication | Baseline (admission day) or no later than 14 days after admission.
  Frequency of renal risk medication prescribed in disagreement to clinical recommendation guidelines based on measured GFR and the choice of eGFR biomarker.
Nutritional status | Baseline (admission day), week 8 and week 16.
  Screening scores for undernutrition with Mini Nutritional Assesment - Short Form, Eating validation scheme, Nutritional Risk Screening-2000
Intestinal microbiome composition | Baseline (admission day), week 8 and week 16 after discharge.
  Composition and changes in the intestinal microbiome.
Body composition | Baseline (admission day), daily through out admission, up to three weeks after admission during kidney function measurement, week 8 and week 16 after discharge.
  Description and changes in body composition, assessed by bioelectric impedance analysis (InBodyS10).
Body composition | Up to three weeks after admission during kidney function measurement
  Assessed by dual x-ray absorptiometry (DXA)

OTHER OUTCOMES:
Number and types of actionable gene variants - Pharmacogenetic test | Baseline (admission day)
  The number of actionable gene variants identified by the pharmacogenetic test
Number and types of recommended therapy changes -Pharmacogenetic test | Baseline (admission day)
  The number of actionable gene variants identified by the pharmacogenetic test
Health economy related to Sub-study 1 | Baseline (admission day), week 8 and week 16 and 1 year after discharge
  Health care costs will be evaluated in regards to changes in quality of life measured by EURO-Qol-5D-5L.

CONTACTS AND LOCATIONS:
Overall Officials: Ove Andersen, MD, PhD, Study Chair — Hvidovre University Hospital; Aino L. Andersen, MSc, Principal Investigator — Hvidovre University Hospital
Locations (1):
- Amager & Hvidovre Hospital, Hvidovre, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Andersen AL, Houlind MB, Nielsen RL, Jorgensen LM, Bengaard AK, Bornaes O, Juul-Larsen HG, Hansen NM, Brochner LD, Hansen RG, Skovlund CAR, Pedersen AML, Beck AM, Pedersen MM, Petersen J, Andersen O. Effectiveness of a multidisciplinary and transitional nutritional intervention compared with standard care on health-related quality of life among acutely admitted medical patients aged >/=65 years with malnutrition or risk of malnutrition: A randomized controlled trial. Clin Nutr ESPEN. 2024 Jun;61:52-62. doi: 10.1016/j.clnesp.2024.02.031. Epub 2024 Mar 13. PMID 38777473
- [Derived] Iversen E, Bengaard AK, Leegaard Andersen A, Tavenier J, Nielsen RL, Juul-Larsen HG, Jorgensen LM, Bornaes O, Jawad BN, Aharaz A, Walls AB, Kallemose T, Dalhoff K, Nehlin JO, Hornum M, Feldt-Rasmussen B, Damgaard M, Andersen O, Houlind MB. Performance of Panel-Estimated GFR Among Hospitalized Older Adults. Am J Kidney Dis. 2023 Dec;82(6):715-724. doi: 10.1053/j.ajkd.2023.05.004. Epub 2023 Jul 28. PMID 37516299